CLINICAL TRIAL: NCT00388349
Title: Gemcitabine and High-dose Chemotherapy Followed by Peripheral Blood Stem Cell Rescue for Relapsed or Resistant Hodgkin's Disease
Brief Title: Gemcitabine and Hodgkin's Disease Chemotherapy Followed by Peripheral Blood Stem Cell Rescue for Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sally Arai, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13511; 1K23AI052413-01A1 (NIH); BMT135 (Other: OnCore)
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Hodgkin Disease; Hodgkin's Lymphoma; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Gemcitabine; Vinorelbine; Carmustine; Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + Autologous HCT (Experimental): Gemcitabine and high-dose chemotherapy followed by peripheral blood stem cell (PBSC) rescue. Chemotherapy includes Gemcitabine + Vinorelbine + Carmustine + Etoposide + Cyclophosphamide.
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine; Drug: Carmustine; Drug: Etoposide; Drug: Cyclophosphamide; Procedure: Autologous HCT

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Vinorelbine
  Other Names: Navelbine
Drug: Carmustine
  Other Names: BCNU
Drug: Etoposide
  Other Names: Vepesid
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar
Procedure: Autologous HCT
  Other Names: Peripheral blood stem cell (PBSC) rescue

SUMMARY:
This is a phase 2 study of gemcitabine + high-dose chemotherapy followed by peripheral blood stem cell (PBSC) rescue for Hodgkin's Disease

DETAILED DESCRIPTION:
To assess the non-hematologic toxicity and determine the phase 2 dose of gemcitabine in combination with vinorelbine followed by carmustine, etoposide and cyclophosphamide and autologous hematopoietic stem cell transplantation [aka peripheral blood stem cell (PBSC)].

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven recurrent or refractory Hodgkin's Disease (Hodgkin's lymphoma) on the basis of excisional biopsy whenever possible.
* Age < 70 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3.
* Phase 1 study component only: 1 or more of the following adverse risk factors

  * Stage IV extranodal disease at relapse "B" symptoms
  * Failure to achieve minimal disease with most recent chemotherapy (single lymph nodes < 2 cm or >75% reduction in a bulky tumor mass and bone marrow involvement < 10%)
  * Progression during induction or salvage therapy
* Phase 2 study component only: No risk factor criteria
* Computerized tomography (CT) scan of the chest, abdomen and pelvis, with assessment of response to last chemotherapy, within 4 weeks of registration. Gallium scan or positron emission tomography (PET) scan confirmation of disease within 4 weeks of registration is highly recommended
* Bone marrow biopsy and cytogenetic analysis within 8 weeks of registration
* Women of child-bearing potential and sexually active males expected to use an accepted and effective method of birth control
* Pretreatment serum bilirubin < 2 x the institutional upper limit of normal (ULN) (within 28 days prior to registration)
* Serum creatinine < 2 x the institutional ULN (within 28 days prior to registration)
* Measured or estimated creatinine clearance > 60 cc/min by the following formula (within 28 days prior to registration):

  * Estimated Creatinine Clearance = (140 age) x WT(kg) x 0.85 (if female) x creatinine (mg/dL)
* Electrocardiogram (ECG) demonstrating no significant abnormalities suggestive of active cardiac disease (within 42 days prior to registration)
* Patients over age 50, who have received chest irradiation or a total of 300 mg/m2 of doxorubicin or with any history of cardiac disease must have a radionuclide ejection fraction (within 42 days prior to registration). If the ejection fraction is 40 to 50%, the patient will have a cardiology consult
* Corrected diffusion capacity > 55%
* Written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Positive HIV antibody test (must be conducted within 42 days of registration)
* No chemotherapy other than corticosteroids should be administered within 2 weeks of the initiation of protocol therapy
* Pregnant
* Breast-feeding
* Requiring therapy for:

  * Coronary artery disease
  * Cardiomyopathy
  * Dysrhythmia, or
  * Congestive heart failure
* Over age 50 and has received chest irradiation or a total of 300 mg/m^2 of doxorubicin
* History of cardiac disease and the ejection fraction is < 40% (radionuclide ejection fraction must be within 42 days of registration)
* Known allergy to etoposide
* History of Grade 3 hemorrhagic cystitis with cyclophosphamide
* History of grade 2 or greater sensory or motor peripheral neuropathy due to prior vinca alkaloid use
* No prior malignancy (EXCEPTION: adequately treated basal cell or squamous cell skin cancer; in situ cervical cancer; or other cancer for which the patients has been disease-free for 5 years). Patients with a prior diagnosis of non-Hodgkin's lymphoma are not eligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2001-09; Primary Completion 2008-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Arai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arai S, Letsinger R, Wong RM, Johnston LJ, Laport GG, Lowsky R, Miklos DB, Shizuru JA, Weng WK, Lavori PW, Blume KG, Negrin RS, Horning SJ. Phase I/II trial of GN-BVC, a gemcitabine and vinorelbine-containing conditioning regimen for autologous hematopoietic cell transplantation in recurrent and refractory hodgkin lymphoma. Biol Blood Marrow Transplant. 2010 Aug;16(8):1145-54. doi: 10.1016/j.bbmt.2010.02.022. Epub 2010 Mar 1. PMID 20197102

RESULTS

PARTICIPANT FLOW:
Groups:
- 1250 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue; 1500 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue: Gemcitabine as administered in combination with vinorelbine, and then followed by high-dose carmustine + etoposide + cyclophosphamide, then autologous peripheral blood stem cell (PBSC) rescue [aka, hematopoietic stem cell transplantation (AHCT)].
Period: Phase I Dose Escalation
Arm/Group | 1250 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue | 1500 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Started | 3 | 4
Completed | 3 | 1
Not Completed | 0 | 3
Not completed — Dose reduction due to DLT | 0 | 3
Period: Phase 2 Dose Expansion
Arm/Group | 1250 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue | 1500 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Started | 139 (Includes the three phase 1 participants who received 1250 mg/m2 gemcitabine (MTD)) | 0 (No participants were treated in Phase 2 at 1500 mg/m2 gemcitabine (MTD exceeded))
Completed (# pts @ 1250 mg/m^2 Gemzar in Phase 2 doesn't include the 4 pts @ 1500 mg/m2 Gemzar in Phase 1.) | 139 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine + High-dose Chemotherapy + PBSC Rescue: Gemcitabine as administered in combination with vinorelbine, and then followed by high-dose carmustine + etoposide + cyclophosphamide, then autologous peripheral blood stem cell (PBSC) rescue [aka, hematopoietic stem cell transplantation (AHCT)].
Arm/Group | Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Number analyzed (Participants) | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 145
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 3
  White | 105
  More than one race | 1
  Unknown or Not Reported | 27

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity of Gemcitabine Due to Non-hematologic Toxicity
Description: Reported as the number of Phase 1 participants by gemcitabine dose that experienced non-hematologic toxicity, ie, drug-related adverse events.
Time Frame: 6 months
Population: 7 patients received 1 of 2 dose levels during the Phase 1 dose-escalation component of the study
Measure: Number; unit: participants
Groups:
- 1250 mg/m2 Gemcitabine + HD Chemo + PBSC Rescue; 1500 mg/m2 Gemcitabine + HD Chemo + PBSC Rescue: Gemcitabine as administered in combination with vinorelbine, and then followed by high-dose carmustine + etoposide + cyclophosphamide, then autologous peripheral blood stem cell (PBSC) rescue [aka, hematopoietic stem cell transplantation (AHCT)].
Arm/Group | 1250 mg/m2 Gemcitabine + HD Chemo + PBSC Rescue | 1500 mg/m2 Gemcitabine + HD Chemo + PBSC Rescue
Number analyzed (Participants) | 3 | 4
participants | 0 | 3

2. Secondary Outcome: Pulmonary Toxicity (BCNU Pneumonitis)
Description: Pulmonary toxicity as assessed by the number of participants that experience BCNU pneumonitis, ie, pneumonitis due to carmustine (BCNU).
Time Frame: 2 years
Population: Patients who completed the study regardless of gemcitabine dose, and had all data points collected.
Measure: Number; unit: participants
Groups:
- Gemcitabine + High-dose Chemotherapy + PBSC Rescue: Gemcitabine (1250 or 1500 mg/m2) administered in combination with vinorelbine, and then followed by high-dose carmustine + etoposide + cyclophosphamide, then autologous peripheral blood stem cell (PBSC) rescue [aka, hematopoietic stem cell transplantation (AHCT)].
Arm/Group | Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Number analyzed (Participants) | 146
participants | 26

3. Secondary Outcome: Overall Survival (OS)
Description: Reports the percentage of participants surviving 6 months after PBSC infusion (transplant).
Time Frame: 2 years
Population: All participants
Measure: Number; unit: percentage of participants
Groups:
- Gemcitabine + High-dose Chemotherapy + PBSC Rescue: Gemcitabine (1250 or 1500 mg/m2) as administered in combination with vinorelbine, and then followed by high-dose carmustine + etoposide + cyclophosphamide, then autologous peripheral blood stem cell (PBSC) rescue [aka, hematopoietic stem cell transplantation (AHCT)].
Arm/Group | Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Number analyzed (Participants) | 146
percentage of participants | 87

4. Secondary Outcome: Relapse Post-transplant
Description: Reports the percentage of participants that experienced relapse post-transplant.
Time Frame: 2 years
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Number analyzed (Participants) | 146
percentage of participants | 29

5. Secondary Outcome: Survival Measures
Description: Reports the survival measures:
  * Freedom from progression (FFP)
  * Event-free survival (EFS)
  * Overall survival (OS)
  EFS and OS were estimated by Kaplan-Meier method
  Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 2 years
Population: Lists the results as included in the publication, which included 92 participants who received the MTD treatment; completed the study; and had all data points collected
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- 1250 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue: Gemcitabine 1250 mg/m2 administered in combination with vinorelbine, and then followed by high-dose carmustine + etoposide + cyclophosphamide, then autologous peripheral blood stem cell (PBSC) rescue [aka, hematopoietic stem cell transplantation (AHCT)].
Arm/Group | 1250 mg/m2 Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Number analyzed (Participants) | 92
percentage of patients
  Freedom from Progression (FFP) | 71 [61 to 81]
  Event-Free Survival (EFS) | 67 [57 to 77]
  Overall Survival (OS) | 83 [75 to 91]

ADVERSE EVENTS:
Time Frame: 2 years
Description: All events reported.
Arm/Group | Gemcitabine + High-dose Chemotherapy + PBSC Rescue
Serious Adverse Events (participants affected / at risk) | 31/146
Other Adverse Events (participants affected / at risk) | 17/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + High-dose Chemotherapy + PBSC Rescue (N=146)
Fever (General disorders) | 2 (2) — persistent fevers included
Constipation (Gastrointestinal disorders) | 3 (3) — Includes severe
Cardiac ischemia (Cardiac disorders) | 1 (1) — myocardial infraction
Ventricular arythmia (Cardiac disorders) | 1 (1) — includes Left ventricular systolic dysfunction
osteomyelitis (Infections and infestations) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Failed to engraft (General disorders) | 1 (1)
Veno-occlusive disease (Cardiac disorders) | 2 (2)
Progressive liver failure (Renal and urinary disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 2 (2)
Allergic reaction (General disorders) | 1 (1)
Relapse (Infections and infestations) | 1 (1)
Intubated (General disorders) | 1 (1)
Multisystem organ failure (General disorders) | 2 (2)
Neutropenia (Infections and infestations) | 1 (1)
Discharge (Blood and lymphatic system disorders) | 1 (1)
Respiratory distress (Cardiac disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1) — including severe
Metabolic abnormalities (Metabolism and nutrition disorders) | 1 (1)
Tachypenic (Cardiac disorders) | 3 (3)
Death (General disorders) | 2 (21)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + High-dose Chemotherapy + PBSC Rescue (N=146)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Arrhythmias (Cardiac disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Friable fascial plane (Blood and lymphatic system disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Candida albicans (Infections and infestations) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
diffusing capacity of the lung for carbon monoxide (DLCO) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated troponin (Blood and lymphatic system disorders) | 1 (1)
Neutropenic fever (Infections and infestations) | 1 (1)
Nodular infiltrates (Blood and lymphatic system disorders) | 1 (1) — Located in right and left lower lobes
Parpneumonic effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes